CLINICAL TRIAL: NCT07176871
Title: Comparing the Alignment Effectiveness of Heat-activated Nickel-titanium (HANT) Versus Conventional Sequences Nickel-titanium (NiTi) Archwires: A Randomized Clinical Trial
Brief Title: Comparing HANT and Conventional NiTi Archwires in Alignment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FOS CTUMP
Record Dates: First submitted 2025-08-30; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Orthodontic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional NiTi AWs (Experimental): even numbers to use conventional NiTi archwire sequences (0.014 NiTi, 0.016 NiTi, 0.016x0.022 NiTi, 0.019x0.025 NiTi, and 0.019x0.025 SS)
  Interventions: Procedure: Archwires
- HANT Aw (Experimental): odd numbers to use HANT arch wires (0.014 NiTi, 0.019x0.025 HANT, and 0.019x0.025 SS).
  Interventions: Procedure: Archwires

INTERVENTIONS:
Procedure: Archwires — All patients were treated with 0.022-inch MBT brackets and sequential NiTi/HANT archwires. A 0.014 NiTi wire was placed initially, followed by monthly archwire changes if no deflection remained. Digital scans were taken from baseline (T0) to 6 months (T6) to measure alignment using Little's irregularity index. Pain was recorded at 24 hours, 3 days, and 1 week with a visual analog scale. CBCT scans before and after alignment assessed root length and alveolar bone changes, with standardized 3D superimpositions ensuring accurate comparisons.

SUMMARY:
This randomized clinical trial evaluated the efficiency of two orthodontic archwire sequences for correcting maxillary anterior crowding. Forty extraction patients (Little's irregularity index: 7-9 mm) were randomly assigned to either a sequence incorporating heat-activated nickel-titanium (HANT) archwires or a conventional NiTi sequence. Digital scans at baseline and monthly intervals up to 6 months assessed alignment changes, while CBCT measured root length and alveolar bone alterations. Pain intensity was recorded using a visual analog scale at 24 hours, 3 days, and 1 week after archwire placement. Statistical significance was set at p ≤ 0.05.

DETAILED DESCRIPTION:
Objective: To compare the clinical efficiency of two sequences of orthodontic wires to correct crowding of the maxillary anterior teeth, one using conventional nickel-titanium (NiTi) archwires and the other utilizing nickel-titanium (NiTi) combined heat-activated nickel-titanium (HANT) archwires in terms of alignment effectiveness, tooth root length, alveolar bone changes, and pain intensity. Methods: Forty patients requiring fixed orthodontic treatment with Little's irregularity index of 7 to 9 mm, who needed first premolar extractions, were recruited. A lottery was conducted for the patients, assigning odd numbers to use HANT archwires (0.014 NiTi, 0.019x0.025 HANT, and 0.019x0.025 SS). (Group 1), and even numbers to use conventional NiTi archwire sequences (0.014 NiTi, 0.016 NiTi, 0.016x0.022 NiTi, 0.019x0.025 NiTi, and 0.019x0.025 SS) (Group 2). Digital scans were taken of the maxilla arch before archwire placement (T0) and at each month (30 days) follow-up leading up to the 6th month (T6). The rate of tooth alignment was measured on digital dental casts by determining Little's irregularity index. The pain experienced by the patient was evaluated 24 hours, 3 days, and 1 week following the placement of the archwire, using a visual analog scale (VAS). Cone beam computed tomographic (CBCT) radiographs of the maxillary anterior teeth were taken before and after alignment to evaluate changes in tooth root length and alveolar bone. Statistical analysis was performed using SPSS software (version 18.0), with significance at p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients with Class I malocclusion on both sides
* aged between 16 and 25 years with permanent dentition
* bilateral extraction of the maxillary first premolar
* maxillary Little's irregularity index between 7-9 mm
* patients with no periodontal disease.

Exclusion Criteria:

* Patients who had previous orthodontic treatment,
* spacing in the maxillary anterior region
* suffer from bleeding disorders, diabetes, bone diseases, periodontal disease, and cancer, as well as those using drugs (such as aspirin, heparin, warfarin, nonsteroidal anti-inflammatory drugs, and glucocorticoids)
* Patients with trauma and facial deformities, smokers, or pregnant were excluded from the study.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Alignment effectiveness | Baseline (T0) and at each month (30 days) follow-up leading up to the 6th month (T6).
  The rate of tooth alignment was measured on digital dental casts by determining Little's irregularity index

SECONDARY OUTCOMES:
Tooth root length | Baseline (T0), After 6 months (T6)
  The change of tooth root length after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No